CLINICAL TRIAL: NCT00545649
Title: Development of Treatments Aiming at Improvement of Function in Patients With Chronic Widespread Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: The Swedish Research Council (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: O687-03-GAU; NCT00569218 (obsolete NCT alias)
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2007-10-17 (Estimated); Status verified 2007-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; chronic pain; physical; exercise; activity; education
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Motor Activity | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Exercise and education
  Interventions: Behavioral: Exercise and education
- 2 (Active Comparator): Education only
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Exercise and education
  Arms: 1
Behavioral: Education
  Arms: 2

SUMMARY:
The study aims to evaluate the effects of adding supervised exercise in supplement to an educational self-management program, and to determine which subgroups would gain effects of the treatment.

DETAILED DESCRIPTION:
164 patients with fibromyalgia and chronic widespread pain were randomized to an exercise-education group or to education-only group. The study period was 20 week. The primary outcome measures comprised the six-minute walk test and the Fibromyalgia Impact Questionnaire. Several other self-administered instruments were included.

ELIGIBILITY:
Inclusion Criteria:

* Women with Fibromyalgia or Chronic widespread pain, aged from 18 to 60 years.

Exclusion Criteria:

* Other somatic or psychiatric disorders, inability to understand Swedish, allergy to chlorine, ongoing treatments or plans to start other treatments during the study period

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2004-05; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Body function (he six-minute walk test) and health status (the Fibromyalgia Impact Questionnaire) | 2004-2007

SECONDARY OUTCOMES:
Self-administered questionnaires assessing distress, stress, quality of life, physical activity, fatigue | 2004-2007

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa Mannerkorpi, Ass prof, Principal Investigator — Göteborg University, Institute of Medicine, Department of Rheumatology and Inflammation Research; Kaisa Mannerkorpi, Ass prof, Principal Investigator — Göteborg University, Institute of Medicine, Department of Rheumtology and Inflammation Research
Locations (3):
- Sweden (3):
  - Alingsas Primary Health Care, Alingsås
  - Göteborg Primary Health Care, Gothenburg
  - Uddevalla Primary Health Care, Uddevalla